CLINICAL TRIAL: NCT06146335
Title: Analysis of Biologic Signatures in Crohn's Patients Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Crohn's & Colitis Foundation of America, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-07026235
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kono-S anastomosis (KSa) (Experimental): Randomized enrollment of preoperative patients undergoing surgical resection for Crohn's ileitis or ileocolitis
  Interventions: Procedure: Kono-S anastomosis (KSa)
- side-to-side anastomosis (SSa) (Active Comparator): Randomized enrollment of preoperative patients undergoing surgical resection for Crohn's ileitis or ileocolitis
  Interventions: Procedure: Side-to-side anastomosis (SSa)

INTERVENTIONS:
Procedure: Kono-S anastomosis (KSa) — antimesenteric functional end-to-end handsewn anastomosis connecting small intestine and colon after surgery
  Arms: Kono-S anastomosis (KSa)
Procedure: Side-to-side anastomosis (SSa) — side-to-side anastomosis connecting small intestine and colon after surgery
  Arms: side-to-side anastomosis (SSa)

SUMMARY:
The purpose of this study is to compare the effect of two procedures - the Kono-S procedure and the side-to-side functional end to end anastomosis - on the microbiome (the bacteria that live in our gut) and on the intestinal immune system. The investigators are hypothesizing that there are differences in the microbiome environment and the immune environment between the two procedural groups.

DETAILED DESCRIPTION:
These are two are different ways to re-connect the intestines after a portion of it is removed during surgery. Patients will be randomly assigned to either be re-connected with a procedure called the Kono-S anastomosis or with a side-to-side anastomosis during their surgery. This study will look at the microbiome and immune environment in the piece of intestine that is removed during surgery. Then, at the follow colonoscopies (3-6 month, 12-18 month, 60 month), biopsies (small pieces of tissue) will be taken near the connection between the small intestine and colon. This will be used to see how the microbiome and immune system in that area changed since the surgery. Genetic tests will be used to measure the microbiome and the levels of immune proteins in the intestines.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Crohn's ileitis/ileocolitis requiring surgical resection OR patients previously enrolled in the "Kono-S anastomosis versus side-to-side functional end anastomosis in the prevention of post-operative recurrence of Crohn's Disease (WC IRB #1303013645)" trial.
2. Patients age 18 years and older.
3. All phenotypes will be included: nonstricturing nonpenetrating (B1), stricturing (B2), and penetrating (B3) according to the Vienna classification.
4. Patients will be included regardless of preoperative medications (untreated, steroids, biologics)

Exclusion Criteria:

1. Patients under 18 years of age.
2. Pregnant patients.
3. Patient does not speak English
4. Patients that may need a different surgical procedure as per the surgeon at the time of intraoperative evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in composition of the microbiome between treatment groups | At the time of the surgery
  Microbiome composition will be measured via an analysis of of 16S rRNA sequencing from tissue samples.
Changes in the immune cell environment between treatment groups | 3-6 month, 12-18 month and 60 month post-surgery endoscopy.
  Immune cell environment in the tissue will be measured by gene expression levels in the tissue sample via bulk RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Michelassi, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No